CLINICAL TRIAL: NCT05527613
Title: Comparison of the Efficacy of a Messaging Application or Verbal Instructions to Improve Oral Hygiene in Patients With Fixed Orthodontic Treatment. Randomized Clinical Trial
Brief Title: Evaluation of the Efficacy of a Messaging Application to Improve Oral Hygiene in Orthodontic Patients.ECA
Acronym: EEMAOHOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Universitaria CIEO (Other)
Responsible Party: Principal Investigator, Claudia Mercedes Ramirez, investigator, Fundación Universitaria CIEO
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Oral hygiene - WhatsApp
Record Dates: First submitted 2022-08-13; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Oral Hygiene; Mobiles Applications
Keywords: Mobiles Applications; Oral Hygiene; Orthodontic Appliances; Fixed; Treatment Outcome

STUDY DESIGN:
Intervention Model Description: consort scheme
Who Masked: Outcomes Assessor
Masking Description: It is not possible to blind the interventions to the patients, nor to the clinicians performing the orthodontic treatment, however the operators, should not know the assignment of the study participants, the processing of the microbiological samples and the statistical advisor will also be blinded, this will be done by means of codes for each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional bracket bonding with instructions by WhatsApp (Experimental): will receive the WhatsApp application, through which oral hygiene reminders will be sent through images and videos with the necessary information, and at the same time they will receive verbal oral hygiene instructions
  Interventions: Other: whatsapp application with oral hygiene reminder for orthodontic patients
- Conventional bracket bonding without instructions by whatsapp (Active Comparator): receive verbal instructions on oral hygiene
  Interventions: Other: whatsapp application with oral hygiene reminder for orthodontic patients

INTERVENTIONS:
Other: whatsapp application with oral hygiene reminder for orthodontic patients — Participants with orthodontics will be randomly assigned to receive the WhatsApp application, through which oral hygiene reminders will be sent using images and videos containing necessary information, and at the same time they will receive verbal instructions on oral hygiene

SUMMARY:
The aim of this article was to compare the efficacy of a messaging application compared to verbal instructions for improving oral hygiene in patients undergoing fixed orthodontic treatment with conventional ligature brackets (MBT technique) over a 3-month period. Randomized clinical trial of two parallel groups with 1:1 allocation ratio. Conducted in the orthodontic postgraduate clinic of the conventional ligation technique (MBT) at the Fundación Universitaria CIEO- UniCIEO, Bogotá, Colombia.

Sixty patients aged 18 to 30 years with periodontal health and active WhatsApp application on smartphone, who started fixed orthodontic treatment with conventional ligation brackets (MBT technique) were included.

Randomization Intervention: all participants received verbal oral hygiene instructions, were randomly assigned by software to the mobile app group (GAM) (n=30) (mean-----DE---- years) that used WhatsApp to reinforce oral hygiene, or to the control group (CG) (n=30) (mean-----DE---- years).

The primary outcome was bacterial plaque level determined with the orthodontic plaque index (OPI) and bleeding on probing (BOP) index measured at three points, after appliance cementation (T0), 1 month later (T1), 2 months later (T2) and 3 months later (T3). Blinding: By two trained operators and blinded to the assignment. The secondary outcome was the identification of microorganisms in the bacterial plaque of the bracket ligation. The data were analyzed by

DETAILED DESCRIPTION:
In this study the researchers are going to recruit patients from the orthodontic clinics with conventional ligation brackets of the MBT technique, from the CIEO - UniCIEO University Foundation; who receive a sequence of archwires, according to the phases of the treatment such as the initial alignment and leveling phase: Nickel - titanium archwires of caliber 0.014, 0.016. Patients entering the study will be randomly assigned to each of the groups; participants in group 1 will receive the WhatsApp application, and at the same time they will receive verbal instructions in oral hygiene; they will be sent reminders, through images and videos with necessary, accurate and instructive information; messages will be sent twice a week for three months. In group 2 the participants will receive verbal instructions given by the researcher on oral hygiene and a video with instructions on the important elements to perform oral hygiene in orthodontic patients. Two indices will also be evaluated: the orthodontic plaque index and the bleeding on probing index.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agree to participate in the study.
* Age from 18 to 30 years
* Patients undergoing orthodontic treatment with fixed appliances using the MBT technique.
* Periodontal health on intact periodontium or diminished periodontium with no history of periodontitis, no presence of bacterial plaque score 0 No plaque deposits on tooth surfaces surrounding the bracket base; according to OPI index, no presence of periodontal pockets, calculus, gingival inflammation and bleeding verified by the periodontist.
* Have cell phone with active WhatsApp application and possibility to connect twice a week, verified by patient interview previously.
* No kinship between participants (affinity/consanguinity)

Exclusion Criteria:

* Systemic history (diabetes, hypertension, poor nutrition), verified by previous patient interview.
* Smokers (smoke 10 cigarettes per day), verified by previous patient interview.
* Pregnancy and lactation.
* Participating in another research or oral health education program.
* Difficulty in speaking or writing Spanish.
* Physical or mental limitation.
* Diagnosis of SARS COV-2.
* Use of mouthwash during the three months of the study.
* Use of additional appliances (lingual arch, transpalatal bar, among others)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-12 (Estimated); Primary Completion 2023-03-25 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in oral hygiene (plaque index (OPI) | the OPI index will be measured over a three-month period
  It will be assessed by the orthodontic plaque index (OPI). The dentition is divided into sextants and the degree of plaque accumulation on each bracket surface (mesial, distal, gingival, incisal/occlusal) and the condition of the adjacent marginal gingivae is assessed. The OPI index is evaluated by four scores or grades; score 0 indicates absence of plaque and inflammation; scores 1 to 3 refer to the severity of plaque accumulations on adjacent brackets and score 4 includes the state of gingival inflammation.
Changes in oral hygiene (bleeding on probing index) | the bleeding on probing index will be measured over a three-month period
  It will be measured by means of the bleeding index according to Loe and Silness. The teeth chosen to apply the gingival index are: 1.6, 2.1, 2.4, 3.6, 4.1, and 4.4, and they are applied in four sites per tooth: distal, vestibular, mesial, and palatal. This means that 24 measurements should be recorded for each patient. The average of the 24 measurements constitutes the Bleeding Index for the whole mouth. At grade 0, there is no bleeding, no bleeding on probing (wait 10 to 30 seconds); at grade 1, there is bleeding, bleeding on probing immediately

SECONDARY OUTCOMES:
microbiological changes (microbiological composition of biofilm) | biofilm sample and microbiological study will be performed at the beginning and in the third month of the study
  The collection of supragingival microbial samples will be collected at the beginning (T0) of the study and at day 90 (T3), after recording the clinical parameters, an explorer will be used as an instrument to remove the elastie or ligature from the bracket and collect the sample from the plaque, which will then be transferred to a transport medium.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Ramirez, Principal Investigator
Locations (1):
- Fundación Universitaria CIEO -UniCIEO, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No